CLINICAL TRIAL: NCT03805971
Title: Probe Based Confocal Laser Endomicroscopy During Thoracoscopy for Pleural Malignancies Diagnosis.
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Olivier Bonhomme, Medical doctor - clinical assistant, University of Liege
Other Study IDs: B707201837069
Record Dates: First submitted 2019-01-13; First posted 2019-01-16 (Actual); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Pleural Carcinomatosis
Keywords: pCLE; confocal laser endomicroscopy; pleural carcinomatosis; mesothelioma; optical biopsies
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Pleural biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient aged more than 18 years admitted for thoracoscopy: Probe based confocal laser endomicroscopy (Mauna kea technologies) will be used, after intravenous fluorescein injection, for every patients admitted for medical thoracoscopy, to study the pleural cavity. Images will be compared with biopsies
  Interventions: Device: Study of the pleural cavity with a confocal laser endomicroscope.

INTERVENTIONS:
Device: Study of the pleural cavity with a confocal laser endomicroscope. — Probe based confocal laser endomicroscope can be introduced through the working chanel of the thoracoscope. this allows the study of the pleural cavity with this new tool.

SUMMARY:
Probe based confocal laser endomicroscopy (pCLE) is a new optical endoscopic technique, generating fluorescent light emission from the tissue of interest and allowing in vivo live imaging at a cellular level ("optical biopsies"). It was first used in gastroenterology and came later to the light in pulmonary medicine and is still an experimental technique. In gastroenterology, this new investigational technique is used in Barret oesophagus, inflammatory bowel disease, pancreas cystic lesions... Nowadays, there are no data concerning usefulness of endomicroscopy in medical thoracoscopy. During thoracoscopy This new tool could help to target biopsies or help clinicians to do the right diagnosis early, allowing rapid therapeutic intervention (talc pleurodesis for example) . Furthermore, some details can be studied only during live imaging as microorganisms or bloodflows. The investigators performed an endomicroscopy to every patient needing a thoracoscopy (no matter the indication) and who agreed to participate. The pCLE features between malignant and benign pleura were compared in order to find specific criteria for malignant infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Every patient refered for a medical thoracoscopy and willing to participate.

Exclusion Criteria:

* < 18 ans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient refered for a medical thoracoscopy and willing to participate.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Bonhomme, MD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonhomme O, Heinen V, Detrembleur N, Corhay JL, Louis R, Duysinx B. Probe-based confocal laser endomicroscopy for pleural malignancies diagnosis. Respirology. 2021 Feb;26(2):188-195. doi: 10.1111/resp.13945. Epub 2020 Oct 1. PMID 33001538

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Aged More Than 18 Years Admitted for Thoracoscopy
Started | 65
Completed | 62
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Patient Aged More Than 18 Years Admitted for Thoracoscopy
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (17.29)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender ratio
  Participants
    Female | 19
    Male | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Thoracoscopy indication [Count of Participants; unit: Participants]
  Talc pleurodesis for recurrent pneumothorax | 8
  Pleural exudation management (mainly lymphocytic) | 46
  Talc pleurodesis for recurrent malignant effusion | 4
  Pleural hyper metabolism on TEP | 2
  Pleural nodularity on CT-scan | 2
Final histological diagnosis [Count of Participants; unit: Participants]
  Normal pleura | 7
  (Sub-)acute pleuritis | 15
  Chronic pleuritis | 13
  Pulmonary adenocarcinoma | 9
  Malignant mesothelioma | 7
  Large cell lymphoma | 2
  Small cell lung carcinoma | 3
  Squamous cell lung carcinoma | 3
  Breast adenocarcinoma | 1
  Urothelial Carcinoma | 1
  Sarcoidosi | 1

OUTCOME MEASURES:

1. Primary Outcome: Pleural Carcinomatosis Identification (Compared to Standard Biopsies). Qualitative Criteria.
Description: Eleven preselected criteria were assessed in their ability to distinguish benign from malignant pleura Qualitative variables are presented in this table
Time Frame: One day.
Measure: Count of Participants; unit: Participants
Groups:
- Benign Pleura: Participants with a benign pleura histological diagnosis.
- Malignant Pleural Infiltrations: Participants with a malignant pleural disease demonstrated by biopsies.
Arm/Group | Benign Pleura | Malignant Pleural Infiltrations
Number analyzed (Participants) | 36 | 26
Participants
  Abnormal tissular architecture: Yes | 8 | 24
  Abnormal tissular architecture: No | 21 | 0
  Abnormal tissular architecture: Not assessable | 7 | 2
  Cellular size homogeneity: Yes | 18 | 7
  Cellular size homogeneity: No | 14 | 16
  Cellular size homogeneity: Not assessable | 4 | 3
  Cellular shape homogeneity: Yes | 18 | 4
  Cellular shape homogeneity: No | 14 | 19
  Cellular shape homogeneity: Not assessable | 4 | 3
  Cellular fluorescence homogeneity: Yes | 28 | 14
  Cellular fluorescence homogeneity: No | 7 | 10
  Cellular fluorescence homogeneity: Not assessable | 1 | 2
  Blood vessels dysplasia: Yes | 8 | 17
  Blood vessels dysplasia: No | 23 | 3
  Blood vessels dysplasia: Not assessable | 5 | 6
  Organized connective tissue: Yes | 11 | 5
  Organized connective tissue: No | 20 | 12
  Organized connective tissue: Not assessable | 5 | 9
  Chia seed sign: Yes | 13 | 0
  Chia seed sign: No | 23 | 26
  Chia seed sign: Not assessable | 0 | 0
Statistical Analysis 1: Comparison: Benign Pleura vs Malignant Pleural Infiltrations; The objective of the test is to assess if the pCLE feature "full chia seed sign" is found statistically more frequently in the "benign pleura group" than in the "malignant pleural infiltrations group"; Test type: Superiority; p = 0.0003, Fisher Exact
Statistical Analysis 2: Comparison: Benign Pleura vs Malignant Pleural Infiltrations; The objective is to assess if the abnormal tissular architecture is significantly more frequently found in the "malignant pleural infiltrations group" than in the "benign pleura group"; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 3: Comparison: Benign Pleura vs Malignant Pleural Infiltrations; The objective is to assess if the pCLE feature "cellular shape homogeneity" is found statistically more frequently in the "benign pleura group" than in the "malignant pleural infiltrations group"; Test type: Superiority; p = 0.0052, Fisher Exact
Statistical Analysis 4: Comparison: Benign Pleura vs Malignant Pleural Infiltrations; The objective is to assess if dysplastic vessels are more frequently found in the "malignant pleural infiltrations group" than in the "benign pleura group"; Test type: Superiority; p < 0.0001, Fisher Exact

2. Primary Outcome: Pleural Carcinomatosis Identification (Compared to Standard Biopsies), Quantitative Criteria.
Description: Eleven preselected pCLE criteria were assessed in their ability to distinguish benign from malignant pleura.
  Here are presented Mean cell size and maximum vascular diameter
Time Frame: One day
Population: Some criteria were not assessable for some patients.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Benign Pleura | Malignant Pleural Infiltrations
Number analyzed (Participants) | 36 | 26
µm
  Mean cell size: number analyzed (Participants) | 29 | 23
  Mean cell size | 21.76 (5.69) | 22.96 (5.16)
  Maximal vascular diameter: number analyzed (Participants) | 27 | 21
  Maximal vascular diameter | 22.72 (9.93) | 27.08 (8.91)

3. Secondary Outcome: Quality of the pCLE Acquisition
Description: The investigators performing the thoracoscopy had to score the pCLE acquisition. Three level of quality were used: Good, Acceptable, Low.
Time Frame: One day
Measure: Count of Participants; unit: Participants
Arm/Group | Benign Pleura | Malignant Pleural Infiltrations
Number analyzed (Participants) | 36 | 26
Participants
  Good | 12 | 8
  Acceptable | 13 | 9
  Low | 11 | 9

4. Primary Outcome: Pleural Carcinomatosis Identification (Compared to Standard Biopsies), Quantitative Criteria.
Description: Eleven preselected pCLE criteria were assessed in their ability to distinguish benign from malignant pleura.
  Quantitative criteria are presented in this table. Here is presented the mean cellular density
Time Frame: One day
Population: Some criteria were not assessable for some patients.
Measure: Mean (Standard Deviation); unit: number of cells/10^4µm^2
Arm/Group | Benign Pleura | Malignant Pleural Infiltrations
Number analyzed (Participants) | 36 | 26
number of cells/10^4µm^2 | 25.42 (8.73) | 22.01 (7.35)

5. Primary Outcome: Pleural Carcinomatosis Identification (Compared to Standard Biopsies), Quantitative Criteria.
Description: Eleven preselected pCLE criteria were assessed in their ability to distinguish benign from malignant pleura.
  Quantitative criteria are presented in this table. Here is presented the vascular density.
Time Frame: One day
Population: Some criteria were not assessable for some patients.
Measure: Mean (Standard Deviation); unit: Vessels/1.13 mm^2 (full optic area)
Arm/Group | Benign Pleura | Malignant Pleural Infiltrations
Number analyzed (Participants) | 36 | 26
Vessels/1.13 mm^2 (full optic area) | 9.81 (7.73) | 6.9 (2.53)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Patient Aged More Than 18 Years Admitted for Thoracoscopy
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT03805971/Prot_SAP_000.pdf